CLINICAL TRIAL: NCT06608225
Title: Prognostic Study of Prostate Cancer Via Dynamic Change of PSA in Peritoneal Drainage Fluid After Radical Prostatectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liu Cheng, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: YLY-PSA
Record Dates: First submitted 2024-09-10; First posted 2024-09-23 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms; Prostate-Specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In this study, biospecimens consist of peritoneal drainage fluid of patients following radical prostatectomy. The fluid is obtained through standard post-operative drainage procedures. The collected samples are analyzed to measure the levels of Prostate-Specific Antigen (PSA) over a designated post-surgical period. The PSA levels in the drainage fluid are dynamically monitored and recorded to assess potential correlations with patient outcomes, recurrence, and metastasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates the prognostic value of dynamic changes in Prostate-Specific Antigen (PSA) levels found in the peritoneal drainage fluid after radical prostatectomy. Prostate cancer is one of the most common cancers in men, and radical prostatectomy is a standard treatment. While PSA levels in the blood are commonly used as a marker for diagnosis, this study focuses on the significance of PSA levels in the prognosis of prostate cancer. The findings may provide insights into improved post-surgical monitoring and more tailored therapeutic strategies for prostate cancer patients.

DETAILED DESCRIPTION:
This study examines the prognostic significance of Prostate-Specific Antigen (PSA) levels in the peritoneal drainage fluid following radical prostatectomy, a common surgical treatment for prostate cancer. PSA is widely used as a biomarker for prostate cancer diagnosis, treatment response, and recurrence monitoring in the blood. However, this research seeks to explore the prognostic value of PSA in the drainage fluid.

The study involves continuous monitoring of PSA levels in the drainage fluid after radical prostatectomy, with the hypothesis that dynamic changes in these levels could serve as an early warning system for potential tumor recurrence, residual disease, or metastasis. The research will correlate these fluid PSA levels with patient outcomes, recurrence rates, and other clinical factors to determine their predictive value.

By investigating this novel source of PSA monitoring, the study aims to reduce invasive tests, enhance post-operative surveillance, and improve early detection of disease recurrence for prostate cancer patients. This research could contribute to refining post-surgical care protocols, offering a new tool for predict long-term outcomes for individuals undergoing radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients treated with radical prostatectomy

Exclusion Criteria:

* 1. Received neoadjuvant endocrine/chemotherapy before surgery;
* 2. Urine leakage after surgery (positive creatinine test of drainage fluid).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include male patients diagnosed with prostate cancer who need radical prostatectomy. Participants must have a preoperative diagnosis confirmed by biopsy and imaging studies. Eligible patients will have an abdominal drainage system in place post-surgery for fluid collection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
PSA Levels in Drainage Fluid | Measured daily for up to 3 days post-surgery.
  Postoperative Prostate-Specific Antigen (PSA) Levels in The Peritoneal Drainage Fluid

CONTACTS AND LOCATIONS:
Overall Officials: Huaqi Zhan, bachelor, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No